CLINICAL TRIAL: NCT04622813
Title: The Effect of Intraoperative Nefopam, Ketoprofen and Paracetamol Combination vs Ketoprofen and Paracetamol Combination on Postoperative Morphine Requirements After Laparoscopic Cholecystectomy: A Randomized, Controlled Trial
Brief Title: Nonopioid Analgesics and Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Sahar Sayyid, Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BIO-2020-0375
Record Dates: First submitted 2020-10-30; First posted 2020-11-10 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Cholecystectomy; Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Nefopam; Ketoprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Patients received sevoflurane-dexmedetomidine-based anesthesia with saline, ketoprofen and paracetamol for postoperative pain control,
  Interventions: Drug: saline infusion, ketoprofen, paracetamol
- Multimodal group (Experimental): patients received sevoflurane-dexmedetomidine-based anesthesia with nefopam, ketoprofen, and paracetamol for postoperative pain control.
  Interventions: Drug: nefopam, ketoprofen, paracetamol

INTERVENTIONS:
Drug: nefopam, ketoprofen, paracetamol — Patients in this group will receive Nefopam and Ketoprofen in addition to the paracetamol intraoperatively prior to the anticipated end of the surgery
  Arms: Multimodal group
Drug: saline infusion, ketoprofen, paracetamol — Patients in this group will receive one placebo infusion (saline infusion) in addition to the ketoprofen and paracetamol intraoperatively prior to the anticipated end of the surgery
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of the addition of nefopam to a multimodal analgesic regimen consisting of ketoprofen and paracetamol during sevoflurane- dexmedetomidine-based anesthesia on postoperative morphine requirements in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Nefopam is a centrally-acting anti-nociceptive compound with supraspinal and spinal sites of action. It inhibits monoamine reuptake, modulates descending serotoninergic pain, and may also interact with a dopaminergic pathway. Because its mechanism of action is distinct from that of other analgesic opioids, nefopam may well have a role in analgesic protocols. The role of nefopam in multimodal analgesia has been extensively investigated in laparoscopic cholecystectomy. However, there is general agreement that more studies are needed to determine the ideal multimodal strategy. No previous study has investigated a combination regimen of the three most commonly prescribed non-opioid analgesics (NOA) (nefopam, ketoprofen, and paracetamol) vs ketoprofen and paracetamol combination during sevoflurane-dexmedetomidine based anesthesia on pain control after laparoscopic cholecystectomy.

The aim of our study is to compare a combination regimen of three NOA (nefopam, ketoprofen, and paracetamol) vs ketoprofen and paracetamol combination during sevoflurane-dexmedetomidine based anesthesia on pain control after laparoscopic cholecystectomy. We will try to demonstrate the benefit with the addition of a third NOA, which is the nefopam, to the double-drug regimen including ketoprofen and paracetamol. Our hypothesis is that this combination regimen of three NOA is associated with less postoperative pain, less opioid consumption, shorter length of post-anesthesia care unit (PACU) stay, and fewer opioid-related adverse effects and postoperative complications compared to the double-drug regimen of ketoprofen and paracetamol.

In this prospective randomized double-blind study, 90 patients aged 18 to 64 years, with American Society of Anesthesiologists (ASA) physical status I and II, will be randomly assigned using a computer-generated random number table to one of two treatment groups. Group A will receive sevoflurane-dexmedetomidine based anesthesia with ketoprofen and paracetamol for postoperative pain control, and group B will receive sevoflurane-dexmedetomidine based anesthesia with nefopam, ketoprofen, and paracetamol for postoperative pain control. The primary outcome measure of this study is total morphine consumption in PACU. Normally distributed data will be summarized as mean ± SD and non-normally distributed data will be summarized as median [interquartile range]. This study would have an impact on our current practice and may help find out the best multimodal analgesic strategy to control postoperative pain after laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Age between 18 and 64 years
* Patients able to give consent

Exclusion Criteria:

* ASA physical status III to V
* History of chronic pain
* Use of an opioid analgesic within 12 hours prior to surgery
* Alcohol or drug abuse
* Chronic opioid intake
* Morbid obesity
* Psychiatric disorder
* Pregnancy or breast-feeding
* Intolerance to NSAIDSs
* Allergy or contraindication to nefopam (acute angle-closure glaucoma, epilepsy, coronary artery disease, prostate adenoma), to morphine or paracetamol (liver failure), to ketoprofen (increased risk of bleeding, stomach or intestinal ulcer, chronic kidney disease) or to dexmedetomidine (uncontrolled hypertension, heart block greater than first degree, or other clinically significant morbidities)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption in the post anesthesia care unit | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  Total morphine doses consumed after the surgery during the post anesthesia care unit stay of the patient

SECONDARY OUTCOMES:
Total fentanyl | Intraoperatively
  Total fentanyl given intraoperatively.
Total morphine | Throughout the patient's stay on the floor
  Total morphine on the floor
Ketoprofen consumption | Throughout the patient's stay on the floor
  Ketoprofen consumption on the floor
Paracetamol consumption | Throughout the patient's stay on the floor
  Paracetamol consumption on the floor
Total morphine consumption at 24 hours after surgery | 24 hours after surgery
  Total morphine doses consumed at 24 hours after surgery
Number of patients receiving morphine in PACU | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  Number of patients receiving morphine in post anesthesia care unit
Number of patients receiving morphine on the floor | Throughout the patient's stay on the floor
  Number of patients receiving morphine on the floor
Number of patients receiving morphine during the first 24 hours after surgery | During the first 24 hours after surgery
  Number of patients receiving morphine during the first 24 hours after surgery
Number of patients receiving ketoprofen on the floor | On the floor
  Number of patients receiving ketoprofen on the floor
Number of patients receiving paracetamol on the floor | On the floor
  Number of patients receiving paracetamol on the floor
NRS pain scores at rest in PACU | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  NRS pain scores at rest in post anesthesia care unit
NRS pain scores at 24 h after surgery | 24 hours after surgery
  NRS pain scores at 24 hours after surgery
sedation scores in PACU | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  sedation scores in post anesthesia care unit
Time to first morphine requirement | From the time of arrival to PACU until discharge
  Time to first morphine requirement
Time to discharge (readiness) from PACU | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  Time to discharge (readiness) from post anesthesia care unit
Nausea and vomiting | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  Incidence and severity of nausea and vomiting
Rescue antiemetics | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  Need for rescue antiemetics
Pruritus | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  Incidence of pruritus
Respiratory depression | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  Incidence of respiratory depression
Urinary retention | Throughout the patient's stay in the recovery room (average of 30 minutes after the surgery)
  Incidence of urinary retention
Tachycardia | Intraoperatively and in PACU
  Episodes of tachycardia
Sweating | Intraoperatively and in PACU
  Episodes of sweating
Quality of recovery | At 24 hours after the surgery
  Quality of recovery at 24 h using the QoR-40
Overall satisfaction score | One month after surgery.
  Overall satisfaction score collected one month after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar Sayyid, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- American University of Beirut Medical center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No